CLINICAL TRIAL: NCT06626854
Title: Prospective, Randomized Study to Assess the Safety and Efficacy of the Novel Noninvasive Hypersound Neuromodulation System in the Treatment of Patients with Chronic Pain of Peripheral Nerve Origin
Brief Title: Treating Chronic Knee Pain with Noninvasive Peripheral Nerve Stimulation Using Novel Interferential RadioFrequencies
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hypersound Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMI01
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Chronic Knee Pain; Chronic Knee Osteoarthritis; Post Surgical Neuropathic Pain
Keywords: rfPNS; Hypersound; Neuroharmonix; Noninvasive PNS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Recipient of Hypersound Therapy
  Interventions: Device: RF-PNS

INTERVENTIONS:
Device: RF-PNS — Noninvasive peripheral nerve stimulator using interferential multi source radio frequency
  Other Names: Noninvasive PNS; Hypersound

SUMMARY:
First, the subject will undergo screening and provide informed consent. Baseline measurements are then taken. The subject remains seated with back support throughout the session. The technician verifies and marks the knee for treatment and wraps an antenna applicator strap around the lower leg near the knee. The device is turned on in test mode to confirm the therapy location, with the subject identifying when they feel a sensation over their pain area. The power threshold for this sensation is recorded. The therapy, which lasts 15 minutes, is delivered at 90% of this threshold to ensure the subject does not feel it. After therapy, post-treatment measurements are taken.

DETAILED DESCRIPTION:
1. Subject will perform screening and informed consent
2. Baseline measurements will be taken
3. Subject will sit in chair with back support throughout duration of the session
4. Knee for treatment will be verified and marked
5. Technician will wrap antenna applicator strap around the lower leg, at the knee
6. Device is turned on and set to test mode to verify therapy location. Subject will verify when they feel a sensation covering their existing chronic knee pain. The power threshold for sensation is recorded.
7. Therapy begins and lasts for 15 minutes, power threshold is set to 90% so that the subject does not feel the therapy
8. At the end of 15 minutes, post-therapy measurements are recorded

ELIGIBILITY:
Inclusion Criteria:

* Pain greater than mid-range using standardized pain inventory (SPI).
* No medication for pain both over-the-counter and by prescription for 24 hours prior to treatment.
* Body mass index (BMI) to be calculated for all participants with limitation for any BMI that is lower than normal. (Target is normal, overweight or obese).
* Age greater than 18.

Exclusion Criteria:

* Existing Peripheral Nerve Stimulator Implant in the lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
VAS | 3 months
  Visual Analog Score Improvement of 50%

SECONDARY OUTCOMES:
Disability | 3 months
  Oswestry disability index improvement of greater than 50%

IPD SHARING:
Plan to Share IPD: No
Staff and research team aren't supported to persist the data